CLINICAL TRIAL: NCT00155337
Title: Photodynamic Therapy for Oral Leukoplakia and Erythroleukoplakia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 9361700753
Record Dates: First submitted 2005-09-08; First posted 2005-09-12 (Estimated); Last update posted 2012-12-21 (Estimated); Status verified 2012-12

CONDITIONS: Oral Leukoplakia
Keywords: leukoplakia; erythroleukoplakia; photodynamic therapy
MeSH Terms: conditions — Leukoplakia, Oral; Leukoplakia | interventions — Photochemotherapy

INTERVENTIONS:
Procedure: photodynamic therapy

SUMMARY:
Photodynamic therapy for oral leukoplakia and erythroleukoplakia

DETAILED DESCRIPTION:
Photodynamic therapy for oral leukoplakia and erythroleukoplakia

ELIGIBILITY:
Inclusion Criteria:

* patients with leukoplakia or erythroleukoplakia

Exclusion Criteria:

* oral cancers

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2004-08; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
End of 8 treatments

SECONDARY OUTCOMES:
Regression of lesions

CONTACTS AND LOCATIONS:
Overall Officials: Chun-Pin Chiang, DMSc, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan